CLINICAL TRIAL: NCT01614626
Title: Alcohol & Zinc Impact on Inflammatory Markers in HIV Disease - Russia ARCH Cohort
Brief Title: Alcohol's Impact on Inflammatory Markers in HIV Disease - Russia ARCH Cohort
Status: Completed | Type: Observational
Sponsor: Boston Medical Center (Other)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Principal Investigator, Jeffrey Samet, Chief, Section of General Internal Medicine, Boston Medical Center
Other Study IDs: H-31200; U01AA020780 (NIH)
Record Dates: First submitted 2012-05-25; First posted 2012-06-08 (Estimated); Last update posted 2020-12-17 (Actual); Status verified 2020-12

CONDITIONS: HIV Infection; Alcohol Use
Keywords: HIV; Alcohol Use; Microbial Translocation; Inflammation; Altered Coagulation; Russia
MeSH Terms: conditions — HIV Infections; Alcohol Drinking; Inflammation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — We are storing serum and plasma for future use, as well as dried blood spots for PEth testing.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The purpose of this study is to assess the longitudinal association between alcohol consumption and biomarkers of microbial translocation (sCD14) and inflammation/altered coagulation (IL-6/D-dimer); to establish a cohort of HIV-infected Russian drinkers; and to establish a sample repository.

DETAILED DESCRIPTION:
Heavy alcohol consumption in an HIV-infected person may accelerate HIV disease progression and end organ disease with one leading explanatory pathway being via enhanced microbial translocation and inflammation/altered coagulation. Heavy alcohol consumption and HIV infection are both causes of microbial translocation, the process by which bacterial products leak across the gastrointestinal membrane with resultant destructive immune activation. Among HIV-infected people, high levels of microbial translocation (as measured by soluble CD14) and inflammation/altered coagulation (as measured by IL-6 and D-dimer) are each associated with an increased risk of death. Of importance, among HIV-infected persons, heavy drinking is also significantly associated with higher levels of D-dimer in cross-sectional studies. Of note, initiation of antiretroviral therapy (ART) is associated with a reduction in D-dimer levels. Yet the following is not known: is there a longitudinal relationship between alcohol consumption and these biomarkers independent of ART?

Thus, as part of the Uganda, Russia, Boston Alcohol Network for Alcohol Research Collaboration on HIV/AIDS (URBAN ARCH)Consortium, the investigators seek to create the Russia ARCH cohort (n=375) from participants of a recently completed NIAAA-funded randomized controlled trial (RCT) of HIV infected Russian heavy drinkers.

The investigators will be collecting blood from participants at baseline, and at 12- and 24-months post enrollment. In addition to collecting and storing blood samples the investigators will be administering surveys to participants at all 3 timepoints. The investigators will conduct phone interviews with participants at 6- and 18-months post enrollment. The investigators will conduct laboratory tests on the stored samples, including measures of microbial translocation (sCD14) and inflammation/altered coagulation (IL-6/D-dimer) and PEth.

This study will clarify the association between alcohol and key biomarkers over time in HIV-infected heavy drinkers. In addition, the investigators will be collecting and storing blood samples from participants in the study to use for the analyses specified and for future studies looking at HIV-infected heavy drinkers.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-70 years old
* HIV-infected
* Provision of contact information for two contacts to assist with follow-up
* Stable address within St. Petersburg or districts within 100 kilometers of St. Petersburg
* Possession of a home or mobile phone
* ART-naive at the time of enrollment

Exclusion Criteria:

* Not fluent in Russian
* Cognitive impairment resulting in inability to provide informed consent

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This is a study of HIV-infected adults who are ART naive at enrollment. Subjects will be recruited from a recently completed NIAAA trial (HERMITAGE; NCT00483483) and from HIV and addiction care sites.
Sampling Method: Non-Probability Sample
Enrollment: 351 (Actual)
Dates: Start 2012-11 (Actual); Primary Completion 2018-04 (Actual); Study Completion 2020-12-15 (Actual)

PRIMARY OUTCOMES:
Microbial translocation as measured by soluble CD14 (sCD14) | Participants will be followed for up to 3 years

SECONDARY OUTCOMES:
Inflammation/altered coagulation as measured by IL-6/D-dimer | Participants will be followed for up to 3 years
Alcohol's association with immunologic aging as measured by flow cytometry | Participants will be followed for up to 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey Samet, MD, MA, MPH, Principal Investigator — Boston Medical Center
Locations (1):
- Pavlov State Medical University, Saint Petersburg, Russia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Related Info — http://www.urbanarch.org